CLINICAL TRIAL: NCT05737134
Title: Mobile Applications Development for Prevention of Sexual Abuse in Elementary School Children by Involving The Roles of Parents and School Teachers in West Java
Brief Title: Mobile Applications Development for Prevention of Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NURS-202212.01
Record Dates: First submitted 2022-12-24; First posted 2023-02-21 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Child Sexual Abuse; Mobile Application

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MA_PESAN APPLICATION (Experimental): The content of MA_PESAN includes an understanding of children, children's rights, sexual understanding, the definition of CSA, forms of CSA, the prevalence of CSA, the impact of CSA, risk factors for the occurrence of CSA, the importance of communication with children, who are the perpetrators/predators of CSA, efforts to prevent CSA. The material is presented in the form of text, images, stop motion videos about the prevention of CSA and videos of the jargon "TANGKIS", songs about "permissible and unacceptable touches", TikTok about "permissible and prohibited touches", and discussion columns. The MA_PESAN intervention was carried out for 9 days.
  Interventions: Other: MA_PESAN MOBILE APPLICATION
- common information from the school (No Intervention): The control group was given intervention according to the procedure at each elementary school. However, information was provided regarding preventing child sexual violence under the procedures usually carried out in each elementary school. The time spent was the same as the intervention group.

INTERVENTIONS:
Other: MA_PESAN MOBILE APPLICATION — The intervention group was given a mobile application consisting of video, and educational material that information was provided regarding the prevention of child sexual abuse.
  Arms: MA_PESAN APPLICATION

SUMMARY:
This interventional study aims to examine the effect of implementing new tools for preventing child sexual abuse (CSA) using a designed digital application for parents/teachers.

The main question of this study is How is the effect of the Mobile Application for Prevention of Sexual Violence in Elementary School-aged Children by Involving the Roles of Parents and School Teachers in West Java on knowledge, attitudes, communication practices, and self-awareness of parents and teachers in West Java.

Two randomized groups of parents will receive or not receive a package of information using a mobile application called MA_PESAN.

The MA_PESAN application is precise and can increase teachers' and parents' knowledge, attitudes, communication practices, and self-awareness about preventing CSA. This application is recommended to be applied in all elementary-level schools.

DETAILED DESCRIPTION:
There is still a lack of knowledge, attitudes, practices, communication skills, and self-awareness among parents and teachers, so education is needed relating to the prevention of CSA. The need to educate parents and teachers is significant because parents are the first teachers of their children in sexual education. Involving parents in educating children about CSA will be effective in encouraging children to use self-protection skills, enabling children to increase safety in the home environment, communication between parents and their children about sexuality, and screening of caregivers. Parents and teachers are the essential sources of providing information to children. The use of media can affect increased knowledge. Several studies on preventing CSA have proven effective in preventing CSA, such as education using discussion methods, pictures, videos, puppets, and sketches.

Education programs regarding the prevention of CSA in schools need to be introduced and taught through schools by involving parents of students at home and teachers at schools, bearing in mind that currently, there is no specific educational program regarding the prevention of CSA in schools. Social media is the dominant communication tool in the 4.0 era. Support can be offered in schools through appropriate methods of preventing CSA due to its broad reach and impact on children's lives. The method is education on the prevention of CSA by using the Mobile Application for Prevention of CSA in Schools (MA_PESAN), which will be developed in this research. The MA_PESAN educational method is education that uses an application intended for parents of students and teachers. The content used in the MA_PESAN material contains material related to the prevention of CSA, the age of children to start being taught CSA prevention, who are the perpetrators/predators of CSA, whether the perpetrators are adults or fellow children, the importance of communication between parents and teachers and children, and eliminating cultural taboos in inform CSA that other studies in the contents of the research material have not carried out.

ELIGIBILITY:
Inclusion Criteria:

* Parents who have elementary school children
* Parents who have an android smartphone and use WhatsApp
* Parents can read
* Parents understand Indonesian
* Have not been exposed to the MA_PESAN educational method

Exclusion Criteria:

* Have physical limitations in using a smartphone
* Parents suffer from illness (are sick)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Knowledge of CSA prevention | 45 days
  Researchers developed this questionnaire. The CSA knowledge instrument contains definitions, forms, determinants, perpetrators of violence, signs and symptoms of victims, impacts, and ways of prevention. The instrument questionnaire consists of 30 questions with multiple-choice options (three answer choices). The correct answer to the positive question is 1, and the wrong answer is 0. Meanwhile, for the negative question, the correct answer is 0, and the wrong answer is 1. Possible scores range from 0-30. The higher the participant's knowledge score, the better their knowledge of CSA prevention.
Attitude toward prevention of Sexual abuse | 45 days
  The researchers developed the instrument. The content of attitude consists of the perception of mothers/teachers of students in grades 5-6 regarding preventing sexual violence. The instrument consists of 13 questions in the form of a Likert scale with a score of 1-4 on a Likert scale. The score for a positive statement is 4 = Strongly Agree; 3=Agreed; 2=Disagree; and 1= Strongly Disagree. Negative questions were changed ('strongly disagree' was coded 4 while 'strongly agree' was coded 1). Possible scores range from 13-52. The higher the participant's attitude score, the more supportive their attitude towards CSA prevention.
Practice of CSA prevention | 45 days
  The authors developed this instrument. The Instrument questionnaire regarding practices on CSA prevention consists of 17 questions. Items for communication practices were measured using a 4-point Likert scale. Contains an attitude statement regarding the prevention of CSA in the form of a Likert scale with a score of 1-4 on a Likert scale. The score for positive statements is 4=Always; 3=often; 2=Rarely; and 1=Never. Negative questions were changed ('never' was coded 4 while 'Always' was coded 1). Possible scores range from 17-68. The higher the participant's communication practice score, the more supportive their communication practice is toward CSA prevention.
Awareness of CSA prevention | 45 days
  The authors developed this instrument. The process of recognizing respondents' thoughts, feelings, and urges is used to guide decision-making regarding preventing sexual violence against children. The instrument questionnaire regarding self-awareness consists of 20 Likert scale questions. Items for self-awareness are measured using a 4-point Likert scale. The attitude scale is: 4=Strongly Agree; 3=Agreed; 2=Disagree; and 1 = Strongly Disagree. Negative questions were changed ('strongly disagree' was coded 4 while 'strongly agree' was coded 1). Possible scores range from 20-80 for self-awareness. The higher the participant's self-awareness score, the higher their self-awareness of CSA prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Henny S Mediani, MNg., PhD, Study Chair — Universitas Padjadjaran
Locations (1):
- University of Padjadjaran, Sumedang, West Java, Indonesia